CLINICAL TRIAL: NCT01474798
Title: A Phase II Open Label Study of the Safety, Pharmacokinetics, and Efficacy of a True Human Anti-Inflammatory Therapeutic Antibody (RA-18C3) in Subjects With Moderate to Severe Acne Vulgaris
Brief Title: Phase II Trial of RA-18C3 in Subjects With Moderate to Severe Acne Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-PT020
Record Dates: First submitted 2011-11-15; First posted 2011-11-18 (Estimated); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Acne Vulgaris
Keywords: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — bermekimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RA-18C3 (Experimental)
  Interventions: Drug: RA-18C3

INTERVENTIONS:
Drug: RA-18C3 — For subjects weighing 27-53 kg: 100 mg (1 ml) administered every three weeks by subcutaneous injection.
  For subjects weighing > 53 kg: 200 mg (2 ml) administered every three weeks by subcutaneous injection.

SUMMARY:
This is a 91-day phase II, open label trial of the true human monoclonal antibody RA-18C3 in subjects with moderate to severe acne vulgaris. Ten (10) subjects will receive RA-18C3 via subcutaneous injection. Subjects will receive injections at Days 0, 21, and 42 for a total of 3 injections. Study drug will be administered under close observation in a facility equipped to handle medical emergencies. Subjects will not be discharged from the facility until at least 1 hour following the injection or 1 hour after their vital signs have stabilized. Safety will be assessed by pre- and post-treatment serial measurements of vital signs, clinical laboratory assessments, and the recording of adverse clinical events.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥ 18
2. Moderate to moderately severe inflammatory acne vulgaris:

   * Investigator's Global Assessment grade of ≥ 3 and,
   * ≥ 15 inflammatory lesions (no more than 6 nodules) and,
   * ≥ 15 non-inflammatory lesions
3. Four week washout period for topical and oral antibiotic treatment
4. Four week washout period for topical retinoids
5. Negative pregnancy test at screening and at specified time points throughout the trial. For subjects with reproductive potential, a willingness to utilize contraception during the study and including 3 months after study completion. Sexually active men must use an accepted method of contraception during the study and including 3 months after study completion.
6. Subjects weighing ≥ 27 kg
7. Signed and dated Institutional Review Board (IRB) approved informed consent before any protocol-specific screening procedures are performed

Exclusion Criteria:

1. A diagnosis of Acne conglobata, acne fulminans, secondary acne, severe nodulocystic acne requiring treatment with isotretinoin, or other dermatologic conditions requiring interfering phototherapy, topical, or systemic treatment.
2. Treatment with any biologicals or investigational agents within the last 4 weeks (or 5 half-lives, whichever is longer).
3. Men with facial hair that would interfere with assessments
4. History of uncontrolled diabetes, unstable ischemic heart disease, active inflammatory bowel disease, active peptic ulcer disease, recent stroke (within 3 months), ongoing congestive heart failure, and any other condition which, in the opinion of the investigator, would put the subject at risk by participation in the protocol.
5. Hemoglobin <10.0 g/dL, or WBC <3.0 x 103/mm3, or platelet count <125 x 103/mm3, or creatinine > 1.5mg/dL, or AST/ALT >2 x ULN, or alkaline phosphatase >2 x ULN
6. Known HIV antibody, hepatitis B surface antigen and/or hepatitis C antibody.
7. History of malignancy within 5 years prior to study entry other than carcinoma in situ of the cervix, or adequately treated, non-metastatic squamous or basal cell carcinoma of the skin.
8. History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies.
9. History of tuberculosis (latent or active) or positive Interferon-gamma release assay (IGRA)
10. Infectious disease:

    * CRP >30 mg/L, fever, or infection requiring treatment with antibiotics within 3 weeks prior to Screening
11. Immunodeficiency
12. Female subjects who are pregnant, planning to become pregnant during the course of the study, or breast-feeding
13. Receipt of a live (attenuated) vaccine within 1 month prior to Screening
14. Major surgery within 28 days prior to Day 0
15. Participation in an investigational drug or device trial within 30 days prior to Screening

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2012-02-29 (Actual); Primary Completion 2012-10-31 (Actual); Study Completion 2012-12-31 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 100 days
  Incidence and type of adverse clinical events

SECONDARY OUTCOMES:
RA-18C3 pharmacokinetics | 70 days
  Serum levels of RA-18C3 will be measured to determine drug half-life, bioavailability, volume of distribution, and area under the curve.
Facial acne lesion count | 56 days
  Change in total facial acne lesion count from day 0 to week 8
Reduction in total acne lesion count, inflammatory and non-inflammatory lesion counts | 56 days
  Percent reduction in total acne lesion count, inflammatory and non-inflammatory lesion counts from day 0 to week 8
Investigator's Global Assessment (IGA) score | 56 days
  Change in Investigator Global Assessment score from baseline to Day 56

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Stecher, MD, Study Director — XBiotech USA, Inc.
Locations (3):
- United States (3):
  - Moy, Fincher, and Chipps Facial Plastics and Dermatology, Beverly Hills, California
  - Meridien Research, St. Petersburg, Florida
  - Austin Dermatology Associates, Austin, Texas